CLINICAL TRIAL: NCT03058484
Title: Short-term Effectiveness of a Community Health Worker Intervention for HIV-infected Pregnant Women in Tanzania to Improve Treatment Adherence and Retention in Care: A Cluster-Randomized Trial
Brief Title: Community Health Workers and Prevention of Mother-to-Child HIV Transmission in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Amref Health Africa (Other); Ministry of Health and Social Welfare, Tanzania (Other Government); International Initiative for Impact Evaluation (Other); Organisation for Public Health Interventions and Development (OPHID) (Unknown)
Responsible Party: Principal Investigator, Sandra McCoy, Assistant Adjunct Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TW7.18; 552553838b402 (Registry Identifier: RIDIE)
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Vertical Transmission of Infectious Disease; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care, i.e. regular clinic services are provided prior to the study.
- Community Health Worker Intervention (Experimental): This arm is a four-part behavioral intervention that includes: 1) formal linkage of CHWs to health facilities; 2) CHW-led antiretroviral therapy (ART) adherence counseling; 3) loss to follow-up tracing by CHWs; and 4) distribution of Action Birth Cards (ABCs), a birth planning tool.
  Interventions: Behavioral: Community Health Worker intervention

INTERVENTIONS:
Behavioral: Community Health Worker intervention — The intervention included four integrated components: 1) formal linkage of CHWs to health facilities; 2) CHW-led antiretroviral therapy (ART) adherence counseling; 3) loss to follow-up tracing by CHWs; and 4) distribution of Action Birth Cards (ABCs), a birth planning tool.
  Arms: Community Health Worker Intervention

SUMMARY:
The investigators implemented and evaluated a pilot program in Shinyanga Region, Tanzania to bring prevention of HIV services to communities using community health workers (CHWs). The intervention aimed to integrate community-based maternal and child health services with HIV prevention, treatment, and care-bridging the gap between women and facility, and enhancing the potential benefits of Option B+. Option B+ is the current World Health Organization recommendation for prevention of mother-to-child transmission, but its success in sub-Saharan Africa may be threatened by overburdened clinics and staff. Consequently, paraprofessionals like CHWs can be key partners in the delivery and/or enhancement of health services in the community.

The study focuses on whether this approach: increases retention in care; improves adherence to antiretrovirals (ARVs); or improves the number of women initiating antiretroviral therapy and the timing of initiation. Investigators hypothesize improvements along primary and secondary outcome indicators in the treatment group. This evaluation helps illuminate both the impact and feasibility of the intervention, and the role that CHWs may play in the elimination of mother-to-child transmission services.

ELIGIBILITY:
Inclusion Criteria:

* Women who were identified in one of the medical registers used for sampling at the facility, were HIV-positive, and had a child born in either the baseline or endline cohort time windows (January and December 2014 or April and October 2015).

Exclusion Criteria:

* Did not have sufficient information to link them across registers

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1830 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Retention in HIV care | 120 days postpartum
  Binary variable taking the value of 1 if the women has had at least one clinic visit in the postpartum period (60-120 days after birth), and zero otherwise.

SECONDARY OUTCOMES:
Adherence to ARVs | Birth to 90 days postpartum
  ART adherence will be measured through a binary variable taking the value of 1 when adherence is at least 95%, and the value of zero otherwise. We measure adherence using the medication possession ratio (MPR), computed as the number of days ARVs are prescribed or dispensed divided by the number of days in the interval. It has been shown to be associated with short-term virologic outcomes.
Timing of ART initiation | ART initiation date, expressed as gestational week of pregnancy, up to 40 weeks
  Defined by gestational week at start of ART, which was computed using standard approaches (i.e., 40 weeks prior to the date of birth or, when available, the expected delivery date based on last menstrual period).
Initiation of ART | Through pregnancy and up to 90 days after birth
  Measured as the number of HIV-infected women in the sample who had any evidence of beginning ART after pregnancy, among women without evidence of treatment prior to pregnancy (women who had initiated ART before the current pregnancy were excluded).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hong SY, Jerger L, Jonas A, Badi A, Cohen S, Nachega JB, Parienti JJ, Tang AM, Wanke C, Terrin N, Pereko D, Blom A, Trotter AB, Jordan MR. Medication possession ratio associated with short-term virologic response in individuals initiating antiretroviral therapy in Namibia. PLoS One. 2013;8(2):e56307. doi: 10.1371/journal.pone.0056307. Epub 2013 Feb 28. PMID 23509605
- [Background] Jaffar S, Amuron B, Foster S, Birungi J, Levin J, Namara G, Nabiryo C, Ndembi N, Kyomuhangi R, Opio A, Bunnell R, Tappero JW, Mermin J, Coutinho A, Grosskurth H; Jinja trial team. Rates of virological failure in patients treated in a home-based versus a facility-based HIV-care model in Jinja, southeast Uganda: a cluster-randomised equivalence trial. Lancet. 2009 Dec 19;374(9707):2080-2089. doi: 10.1016/S0140-6736(09)61674-3. Epub 2009 Nov 24. PMID 19939445
- [Background] Geldsetzer P, Yapa HM, Vaikath M, Ogbuoji O, Fox MP, Essajee SM, Negussie EK, Barnighausen T. A systematic review of interventions to improve postpartum retention of women in PMTCT and ART care. J Int AIDS Soc. 2016 Apr 25;19(1):20679. doi: 10.7448/IAS.19.1.20679. eCollection 2016. PMID 27118443
- [Background] Mwai GW, Mburu G, Torpey K, Frost P, Ford N, Seeley J. Role and outcomes of community health workers in HIV care in sub-Saharan Africa: a systematic review. J Int AIDS Soc. 2013 Sep 10;16(1):18586. doi: 10.7448/IAS.16.1.18586. PMID 24029015
- [Background] Anyangwe SC, Mtonga C. Inequities in the global health workforce: the greatest impediment to health in sub-Saharan Africa. Int J Environ Res Public Health. 2007 Jun;4(2):93-100. doi: 10.3390/ijerph2007040002. PMID 17617671
- [Derived] Nance N, Pendo P, Masanja J, Ngilangwa DP, Webb K, Noronha R, McCoy SI. Short-term effectiveness of a community health worker intervention for HIV-infected pregnant women in Tanzania to improve treatment adherence and retention in care: A cluster-randomized trial. PLoS One. 2017 Aug 31;12(8):e0181919. doi: 10.1371/journal.pone.0181919. eCollection 2017. PMID 28859083